CLINICAL TRIAL: NCT00553852
Title: Evaluation of GH/IGF-I Axis and of Replacement GH Therapy After Bariatric Surgery in Patients With Very Severe Obesity: Relationships With Body Composition
Brief Title: Replacement GH Therapy After Bariatric Surgery in Patients With Very Severe Obesity
Acronym: GH&LASGB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Annamaria Colao, Department of Molecular and Clinical Endocrinology and Oncology University Federico II of Naples
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeuroendoUnit-5
Record Dates: First submitted 2007-10-31; First posted 2007-11-06 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Obesity; GHD
Keywords: Very Severe Obesity; Body Composition; GH deficiency; IGF-I; LASGB; GH therapy
MeSH Terms: conditions — Obesity; Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The clinical examination will determine anthropometric indexes (weight, height, BMI, waist circumference). The biochemical evaluation will include the measurement of lipid profile, fasting plasma glucose and insulin, liver test function, FT3, FT4, GHRH + Arginine test to detect GHD, plasma IGF-I levels. The instrumental evaluation will include DEXA Total Body and bioimpedance analysis to determine body composition, and liver ultrasounds.
  Interventions: Drug: Recombinant GH Saizen (Merck-Serono)
- 2 (Placebo Comparator): PHASE II: In the medical treatment protocol very severe obese patients with persistent GHD after LASGB will be inclosed. Starting from 15-day, GHD patients were re-evaluated by GHRH + Arginine test. After evaluation, the patients with persistent GHD will be randomized to be treated with Recombinant GH replacement therapy (Group A: Recombinant GH replacement therapy at the initial dose 0.15-0.30 mg/die; dose adjustment will be made according to IGF-I levels; Group B: no GH treatment).
  Interventions: Drug: Recombinant GH Saizen (Merck-Serono)

INTERVENTIONS:
Drug: Recombinant GH Saizen (Merck-Serono) — Treatment will start at the initial dose 0.15-0.30 mg/day; dose adjustment will be performed according to IGF-I levels. The duration of medical treatment is 6 months.

SUMMARY:
Obesity and obesity-related diseases have reached epidemic proportions in Western countries (1-3). Laparoscopic-adjustable silicone gastric banding (LASGB) is a purely restrictive operation that determine effective weight loss without inducing malabsorption (4-6). However, also after LASGB body weight loss is almost invariably associated with Free Fat Mass (FFM) loss, and the relevance of the FFM contribution to total energy expenditure is well-known (7-8). Different endocrine axes are reported to affect FFM. We previously reported that low levels of DHEA-S, an adrenal steroid with controversial anti-adipogenic and anti-atherogenic effects, are increased after the massive and sustainable weight loss induced by LASGB in severely obese premenopausal women and correlated with the higher post-operative FFM (9-10). It is also well known that GH/IGF-I axis exerts relevant effects on FFM and that reduced GH levels might increase Fat Mass (FM) and reduce FFM (11,12). Morbidly obese patients have a reduced GH secretion, generally reversible after weight loss (13-14). In a recent study currently in press, we reported that a persistent deficiency in the GH/IGF-I axis in very obese females is associated to lower decrease in FM after LASGB. Low IGF-I plasma levels have also been reported to be independent prognostic factors of liver steatosis and non-alcoholic steatohepatitis in morbidly obese patients (15) and ultrasound- measured hepatic left lobe volume might represent a reliable tool for the evaluation of liver involvement in obesity (16). GH deficiency (GHD) in adult patients is associated with an increase in FM and a parallel decrease in FFM (17). The severity of GDH is correlated to cardiovascular risk, body composition abnormalities and bone loss, and decreased left ventricular ejection fraction (18-20). GH therapy has been demonstrated to be effective in normalizing body composition, with beneficial effects up to a 2-years follow-up period (21-24). GH therapy has also been reported to be effective in sparing FFM during weight loss in obese patients and metabolic syndrome (25,26). However, these studies have some limitations due to the duration of the treatment and the lack of a preliminary evaluation of the GH/IGF-I axis secretory status in obese patients before the GH therapy. At present there are no data on the evaluation of the GH/IGF-I status before and after bariatric surgery and the effectiveness of recombinant GH treatment in very severe obese patients.

DETAILED DESCRIPTION:
The objectives of the study are:

1. To evaluate the GH/GF-I status is correlation with body composition in very severe obese patients. IGF-I levels were classified as deficient when the standard deviation score from the mean was <-2 for age and gender.
2. To evaluate the efficacy of a medical treatment with recombinant GH replacement therapy in very severe obese patients after LASGB on the Fat mass (%), free fat mass (%), percent decrease of fat mass. In line with GHD diagnosis, obese patients with persistent GHD after bariatric surgery will be randomized to be treated with or without recombinant GH therapy with replacement doses, in addition to the controlled trial of dietary management, as routinely performed after LASGB.

Study protocol The study protocol includes two different arms: a correlation observational longitudinal open study (Phase I), and a treatment study (Phase II).

PHASE I: In the correlation study a clinical, biochemical and instrumental evaluation will be performed in 20-30 patients with very severe obesity (grade III) with GHD followed-up in a multi-disciplinary approach at the Unit of Endocrinology of the Departments of Molecular and Clinical Endocrinology and Oncology and at the Physiology Nutrition Unit of the Department of Neuroscience and the Department of Surgery of "S. Giovanni Bosco" Hospital of Naples, according to the current criteria of the National Institute of Health (27). The clinical examination will focus on the GH/IGF-I status effects on body composition changes before and after LASGB. The clinical examination will determine anthropometric indexes (weight, height, BMI, waist circumference). The biochemical evaluation will include the measurement of lipid profile, fasting plasma glucose and insulin, liver test function, FT3, FT4, GHRH + Arginine test to detect GHD, plasma IGF-I levels. The instrumental evaluation will include DEXA Total Body and bioimpedance analysis to determine body composition, and liver ultrasounds.

PHASE II: In the medical treatment protocol very severe obese patients with persistent GHD after LASGB will be inclosed. Starting from 15-day, GHD patients were re-evaluated by GHRH + Arginine test. After evaluation, the patients with persistent GHD will be randomized to be treated with Recombinant GH replacement therapy (Group A: Recombinant GH replacement therapy at the initial dose 0.15-0.30 mg/die; dose adjustment will be made according to IGF-I levels; Group B: no GH treatment). In both subgroups, the diet will arranged to fit an energy intake of 5.7 MJ/day (55% carbohydrate, 25% fat, 20% protein, 30 g fiber) and a moderate-intensity activity (brisk walking for 30-45 min/day) will be encouraged.

The evaluation of medical treatment efficacy will be based on the analysis of changes in anthropometric indexes, IGF-I levels, liver function test, body composition assessed by DEXA Total Body and bioimpedance analysis, liver ultrasounds. At 3 and 6 months, the patients of both subgroups A and B will be clinically re-evaluated, plasma samples for metabolic, liver function tests, and endocrine profile will be obtained, body composition and liver ultrasounds will be determined. At the end of the 6-months period of treatment and observation, the GH response to a subsequent GHRH + Arginine will be re-tested to confirm or to exclude GHD. All the patients with persistent GHD will continue recombinant GH therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50 yrs
* Normal glucose tolerance during standard oral glucose tolerance test (OGTT)
* Inclusion criteria for bariatric surgery proposed by the 1991 National Institutes of Health Consensus Development Panel Report.

Exclusion Criteria:

* Liver or renal failure, cancer, acute or chronic inflammatory diseases
* Chronic treatment with any type of medications
* organic pituitary deficiency
* Bulimia Nervosa of the DSM-IV
* Ulcers or malignancies excluded by oesophagus-gastro-duodenoscopy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Fat mass (%), free fat mass (%), percent decrease of fat mass. | 6 months

SECONDARY OUTCOMES:
Lipid profile | 6 months
Fasting plasma glucose and insulin | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Colao, MD, PhD, Principal Investigator — Department of Molecular and Clinical Endocrinology and Oncology Federico II University of Naples
Locations (1):
- Department of Molecular and Clinical Endocrinology and Oncology Federico II University, Naples, Italy

REFERENCES:
- [Background] Groves T. Pandemic obesity in Europe. BMJ. 2006 Nov 25;333(7578):1081. doi: 10.1136/bmj.39038.449769.BE. Epub 2006 Nov 17. PMID 17114210
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Background] Renehan AG, Frystyk J, Flyvbjerg A. Obesity and cancer risk: the role of the insulin-IGF axis. Trends Endocrinol Metab. 2006 Oct;17(8):328-36. doi: 10.1016/j.tem.2006.08.006. Epub 2006 Sep 7. PMID 16956771
- [Background] DeMaria EJ. Bariatric surgery for morbid obesity. N Engl J Med. 2007 May 24;356(21):2176-83. doi: 10.1056/NEJMct067019. No abstract available. PMID 17522401
- [Background] Kuzmak LI. A Review of Seven Years' Experience with Silicone Gastric Banding. Obes Surg. 1991 Dec;1(4):403-408. doi: 10.1381/096089291765560809. PMID 10775942
- [Background] Angrisani L, Lorenzo M, Esposito G, Romano G, Puzziello A, Belfiore A, Santoro T, Roina G, Petito A, Falconi C, Tesauro B. Laparoscopic adjustable silicone gastric banding: preliminary results of the University of Naples experience. Obes Surg. 1997 Feb;7(1):19-21. doi: 10.1381/096089297765556178. PMID 9730532
- [Background] Ravussin E, Burnand B, Schutz Y, Jequier E. Energy expenditure before and during energy restriction in obese patients. Am J Clin Nutr. 1985 Apr;41(4):753-9. doi: 10.1093/ajcn/41.4.753. PMID 3984927
- [Background] Sergi G, Lupoli L, Busetto L, Volpato S, Coin A, Bertani R, Calliari I, Berton A, Enzi G. Changes in fluid compartments and body composition in obese women after weight loss induced by gastric banding. Ann Nutr Metab. 2003;47(3-4):152-7. doi: 10.1159/000070038. PMID 12743467
- [Background] Savastano S, Valentino R, Belfiore A, De Luca N, de Alteriis A, Orio F Jr, Palomba S, Villani AM, Falconi C, Lupoli G, Lombardi G. Early carotid atherosclerosis in normotensive severe obese premenopausal women with low DHEA(S). J Endocrinol Invest. 2003 Mar;26(3):236-43. doi: 10.1007/BF03345163. PMID 12809174
- [Background] Savastano S, Belfiore A, Guida B, Angrisani L, Orio F Jr, Cascella T, Milone F, Micanti F, Saldalamacchia G, Lombardi G, Colao A. Role of dehydroepiandrosterone sulfate levels on body composition after laparoscopic adjustable gastric banding in pre-menopausal morbidly obese women. J Endocrinol Invest. 2005 Jun;28(6):509-15. doi: 10.1007/BF03347238. PMID 16117191
- [Background] Richelsen B, Pedersen SB, Kristensen K, Borglum JD, Norrelund H, Christiansen JS, Jorgensen JO. Regulation of lipoprotein lipase and hormone-sensitive lipase activity and gene expression in adipose and muscle tissue by growth hormone treatment during weight loss in obese patients. Metabolism. 2000 Jul;49(7):906-11. doi: 10.1053/meta.2000.6738. PMID 10910003
- [Background] Umpleby AM, Russell-Jones DL. The hormonal control of protein metabolism. Baillieres Clin Endocrinol Metab. 1996 Oct;10(4):551-70. doi: 10.1016/s0950-351x(96)80711-7. PMID 9022951
- [Background] Maccario M, Grottoli S, Procopio M, Oleandri SE, Rossetto R, Gauna C, Arvat E, Ghigo E. The GH/IGF-I axis in obesity: influence of neuro-endocrine and metabolic factors. Int J Obes Relat Metab Disord. 2000 Jun;24 Suppl 2:S96-9. doi: 10.1038/sj.ijo.0801289. PMID 10997620
- [Background] Garcia-Galiano D, Sanchez-Garrido MA, Espejo I, Montero JL, Costan G, Marchal T, Membrives A, Gallardo-Valverde JM, Munoz-Castaneda JR, Arevalo E, De la Mata M, Muntane J. IL-6 and IGF-1 are independent prognostic factors of liver steatosis and non-alcoholic steatohepatitis in morbidly obese patients. Obes Surg. 2007 Apr;17(4):493-503. doi: 10.1007/s11695-007-9087-1. PMID 17608262
- [Background] Santini F, Giannetti M, Mazzeo S, Fierabracci P, Scartabelli G, Marsili A, Valeriano R, Pucci A, Anselmino M, Zampa V, Vitti P, Pinchera A. Ultrasonographic evaluation of liver volume and the metabolic syndrome in obese women. J Endocrinol Invest. 2007 Feb;30(2):104-10. doi: 10.1007/BF03347407. PMID 17392599
- [Background] Molitch ME, Clemmons DR, Malozowski S, Merriam GR, Shalet SM, Vance ML; Endocrine Society's Clinical Guidelines Subcommittee; Stephens PA. Evaluation and treatment of adult growth hormone deficiency: an Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2006 May;91(5):1621-34. doi: 10.1210/jc.2005-2227. Epub 2006 Apr 24. PMID 16636129
- [Background] Colao A, Cerbone G, Pivonello R, Aimaretti G, Loche S, Di Somma C, Faggiano A, Corneli G, Ghigo E, Lombardi G. The growth hormone (GH) response to the arginine plus GH-releasing hormone test is correlated to the severity of lipid profile abnormalities in adult patients with GH deficiency. J Clin Endocrinol Metab. 1999 Apr;84(4):1277-82. doi: 10.1210/jcem.84.4.5605. PMID 10199767
- [Background] Colao A, Di Somma C, Pivonello R, Loche S, Aimaretti G, Cerbone G, Faggiano A, Corneli G, Ghigo E, Lombardi G. Bone loss is correlated to the severity of growth hormone deficiency in adult patients with hypopituitarism. J Clin Endocrinol Metab. 1999 Jun;84(6):1919-24. doi: 10.1210/jcem.84.6.5742. PMID 10372687
- [Background] Colao A, Di Somma C, Cuocolo A, Filippella M, Rota F, Acampa W, Savastano S, Salvatore M, Lombardi G. The severity of growth hormone deficiency correlates with the severity of cardiac impairment in 100 adult patients with hypopituitarism: an observational, case-control study. J Clin Endocrinol Metab. 2004 Dec;89(12):5998-6004. doi: 10.1210/jc.2004-1042. PMID 15579750
- [Background] Salomon F, Cuneo RC, Hesp R, Sonksen PH. The effects of treatment with recombinant human growth hormone on body composition and metabolism in adults with growth hormone deficiency. N Engl J Med. 1989 Dec 28;321(26):1797-803. doi: 10.1056/NEJM198912283212605. PMID 2687691
- [Background] Vance ML, Mauras N. Growth hormone therapy in adults and children. N Engl J Med. 1999 Oct 14;341(16):1206-16. doi: 10.1056/NEJM199910143411607. No abstract available. PMID 10519899
- [Background] Amato G, Mazziotti G, Di Somma C, Lalli E, De Felice G, Conte M, Rotondi M, Pietrosante M, Lombardi G, Bellastella A, Carella C, Colao A. Recombinant growth hormone (GH) therapy in GH-deficient adults: a long-term controlled study on daily versus thrice weekly injections. J Clin Endocrinol Metab. 2000 Oct;85(10):3720-5. doi: 10.1210/jcem.85.10.6881. PMID 11061530
- [Background] Johannsson G, Marin P, Lonn L, Ottosson M, Stenlof K, Bjorntorp P, Sjostrom L, Bengtsson BA. Growth hormone treatment of abdominally obese men reduces abdominal fat mass, improves glucose and lipoprotein metabolism, and reduces diastolic blood pressure. J Clin Endocrinol Metab. 1997 Mar;82(3):727-34. doi: 10.1210/jcem.82.3.3809. PMID 9062473
- [Background] Albert SG, Mooradian AD. Low-dose recombinant human growth hormone as adjuvant therapy to lifestyle modifications in the management of obesity. J Clin Endocrinol Metab. 2004 Feb;89(2):695-701. doi: 10.1210/jc.2003-031264. PMID 14764783
- [Background] NIH conference. Gastrointestinal surgery for severe obesity. Consensus Development Conference Panel. Ann Intern Med. 1991 Dec 15;115(12):956-61. PMID 1952493
- [Result] Savastano S, Di Somma C, Belfiore A, Guida B, Orio F Jr, Rota F, Savanelli MC, Cascella T, Mentone A, Angrisani L, Lombardi G, Colao A. Growth hormone status in morbidly obese subjects and correlation with body composition. J Endocrinol Invest. 2006 Jun;29(6):536-43. doi: 10.1007/BF03344144. PMID 16840832
- [Derived] Savastano S, Di Somma C, Angrisani L, Orio F, Longobardi S, Lombardi G, Colao A. Growth hormone treatment prevents loss of lean mass after bariatric surgery in morbidly obese patients: results of a pilot, open, prospective, randomized, controlled study. J Clin Endocrinol Metab. 2009 Mar;94(3):817-26. doi: 10.1210/jc.2008-1476. Epub 2008 Dec 9. PMID 19066295